CLINICAL TRIAL: NCT01944553
Title: A Prospective Study on the Feasibility of Pedicle Screw Placement in the Lumbar Level With a New Robotic-assisted System
Brief Title: Robotic-assisted Pedicule Screw Placement
Acronym: ARASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Medtech S.A.S (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF 9180; 2013-A00749-36 (Other: ID-RCB)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Lumbar Degenerative Spinal Disease
Keywords: Spine; Accurancy; Robotic; Screw placement; Degenerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prospective (Experimental): Single Arm
  Interventions: Device: The ROSA™ robot

INTERVENTIONS:
Device: The ROSA™ robot — The ROSA™ robot can assist in identifying the pedicle entry point and in controlling the screw trajectory through a system of continuous monitoring of patient motion. This process strengthens the accuracy of pedicle screws implantation.
  Stabilisation in treatment for spine degenerative disease

SUMMARY:
The main objective of the study is to evaluate the feasibility of using the robotic assisted device ROSA™ for pedicle screws placement. This device is currently used in cranial neurosurgery but its applications can be extended to other fields, such as spinal surgery. In the future, the use of ROSA™ in pedicle screw placement could increase the accuracy and safety of surgery for the patient.

DETAILED DESCRIPTION:
The medical device subject of this research is the surgical robot ROSA™ designed for cranial surgery, and used here in another application, spinal surgery - more specifically for the placement of pedicle screws.

It is intended for spine surgeons to treat diseases requiring the placement of pedicle screws through posterior open surgery approach or minimally invasive surgery.

The system allows the precise guidance of instruments as defined by the surgeon on patient radiological images. The expected performance is a good rate of pedicle screws placement, increasing the performance observed with the conventional method. This system can be transported from one operating room to another, and stored in a storage room.

It interfaces with the most common intra -operative surgical imaging systems (mobile C-arms available at Montpellier University Hospital). Further versions of the device will enable the use of 3D intra-operative imaging systems such as the O-arm from Medtronic.

The main objective of the study is to evaluate the feasibility of using the robot ROSA™ for pedicle screws placement. In this study, the robot will be used with an open surgery approach, which is a first step in demonstrating the potential of the robot.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from lumbar back pain for more than 3 months
* Consent signed

Exclusion Criteria:

* pregnant patient
* patient nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
accurancy of pedicle screw placement | during the surgery
  The main objective of the study is to evaluate the feasibility of the robot ROSA in the pedicle screw placement anf for obtaining a CE mark for this application.The expected performance are a "good rate positioning" of pedicle screws better than the performance observed in conventional surgery.

SECONDARY OUTCOMES:
operative time / irradiation doses | During the surgery
  The secondary outcome of the study is to evaluate the operative time and the irradiation doses during the surgery with this medical device.

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier Hospital, Montpellier, France